CLINICAL TRIAL: NCT02761642
Title: Multicenter Study for the Evaluation of Efficacy and Safety of NeoRecormon® Therapy Administered as 30000 IU Subcutaneously in Anemic Patients With Breast Cancer Treated With Chemotherapy
Brief Title: A Study to Evaluate Efficacy and Safety of Epoetin Beta (NeoRecormon®) in Anemic Participants With Breast Cancer Undergoing Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML17503
Record Dates: First submitted 2016-05-03; First posted 2016-05-04 (Estimated); Results first posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — epoetin beta

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Epoetin Beta (Experimental): Anemic breast cancer participants will receive epoetin beta treatment for 12 weeks.
  Interventions: Drug: Epoetin Beta

INTERVENTIONS:
Drug: Epoetin Beta — All participants will receive epoetin beta at a dose of 30000 International Units (IU) as SC injection once every week for a total of 12 weeks. Adjustments in the dose will be implemented based on the participant's blood hemoglobin levels.
  Other Names: NeoRecormon

SUMMARY:
This study will evaluate the efficacy and safety of subcutaneous (SC) epoetin beta in anemic participants with breast cancer undergoing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult female participants with histological diagnosis of breast cancer
* Any type of chemotherapy planned for greater than or equal to (>/=) 9 weeks
* Hemoglobin level less than (<) 11 grams per deciliter (g/dL)
* Participants able to receive iron supplement, if necessary

Exclusion Criteria:

* Known or suspected contraindications to epoetin beta
* Pregnancy or lactation period
* Diagnosis of anemia only due to iron-deficiency
* Diagnosis of thalasemic syndromes
* Epilepsy and/or cerebral metastasis
* Blood transfusion or treatment with any erythropoietic factor within 4 weeks before study start

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2004-02-29 (Actual); Primary Completion 2007-03-31 (Actual); Study Completion 2007-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (26):
- Italy (26):
  - Arezzo
  - Ascoli Piceno
  - Bussolengo VR
  - Busto Arsizio
  - Casale Monferrato
  - Catania
  - Catanzaro
  - Chieti
  - Cuneo
  - Fano
  - Florence
  - Frosinone
  - Genova
  - Macerata
  - Messina
  - Monza
  - Napoli
  - Nocera Inferiore
  - Pavia
  - Pisa
  - Pordenone
  - Roma
  - Sassari
  - Torino
  - Vecchiazzano
  - Vittorio Veneto

RESULTS

PARTICIPANT FLOW:
Groups:
- Epoetin Beta: Anemic breast cancer participants received epoetin beta (NeoRecormon®) at a dose of 30000 International Units (IU) as subcutaneous (SC) injection once every week for a total of 12 weeks. Adjustments in the dose were implemented based on the participant's blood hemoglobin levels.
Period: Overall Study
Arm/Group | Epoetin Beta
Started | 200
Treated | 197
Completed | 130
Not Completed | 70
Not completed — Did not Receive Study Treatment | 3
Not completed — Adverse Event | 13
Not completed — Withdrawal by Subject | 2
Not completed — Non-compliant | 7
Not completed — Death | 3
Not completed — Lack of Efficacy | 20
Not completed — Physician Decision | 1
Not completed — Reason Unspecified | 21

BASELINE CHARACTERISTICS:
Population: Safety population: included all enrolled participants who received at least 1 dose of study drug.
Arm/Group | Epoetin Beta
Number analyzed (Participants) | 197
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response to Treatment Based on Hemoglobin Levels
Description: Response was defined as increase of hemoglobin levels by at least 2 grams per deciliter (g/dL) as compared to baseline or the achievement of hemoglobin level of 12 g/dL after 12 weeks of treatment in the absence of red blood cells transfusion.
Time Frame: Week 12
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Epoetin Beta
Number analyzed (Participants) | 197
percentage of participants | 46.2 [38.2 to 54.3]

2. Secondary Outcome: Change From Baseline in Hemoglobin Levels After 12 Weeks of Study Treatment in Participants According to the Hemoglobin Level at Baseline
Description: Participants were distributed into 2 subgroups. One subgroup contained participants who had hemoglobin (Hb) level less than (<) 10 g/dL and other subgroup contained participants who had hemoglobin level greater than or equal to (≥) 10 g/dL but <11 g/dL (10≤ Hb <11 g/dL).
Time Frame: Baseline, Week 12
Population: Safety population. Here, "Number Analyzed" represents number of participants evaluable for the specified category.
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Epoetin Beta
Number analyzed (Participants) | 197
g/dL
  Baseline; Hb <10 g/dL: number analyzed (Participants) | 89
  Baseline; Hb <10 g/dL | 9.4 [9.3 to 9.5]
  Baseline; 10≤ Hb <11 g/dL: number analyzed (Participants) | 108
  Baseline; 10≤ Hb <11 g/dL | 10.5 [10.4 to 10.6]
  Change at Week 12; Hb <10 g/dL: number analyzed (Participants) | 89
  Change at Week 12; Hb <10 g/dL | 2.1 [1.8 to 2.4]
  Change at Week 12; 10≤ Hb <11 g/dL: number analyzed (Participants) | 108
  Change at Week 12; 10≤ Hb <11 g/dL | 1.1 [0.9 to 1.3]

3. Secondary Outcome: Change From Baseline in Hemoglobin Levels After 12 Weeks of Study Treatment in Participants According to Chemotherapy at Baseline
Description: Participants were distributed into 3 subgroups. First subgroup contained participants who received adjuvant chemotherapy. Second subgroup contained participants who received metastatic 1st or 2nd line chemotherapy. Third subgroup contained participants who received metastatic 3rd line chemotherapy.
Time Frame: Baseline, Week 12
Population: Safety population. Here, "Number Analyzed" represents number of participants evaluable for the specified category.
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Epoetin Beta
Number analyzed (Participants) | 197
g/dL
  Baseline; Adjuvant Chemotherapy: number analyzed (Participants) | 70
  Baseline; Adjuvant Chemotherapy | 10.2 [10.0 to 10.3]
  Baseline; Metastatic 1st or 2nd Line: number analyzed (Participants) | 92
  Baseline; Metastatic 1st or 2nd Line | 9.8 [9.6 to 9.9]
  Baseline; Metastatic 3rd Line: number analyzed (Participants) | 35
  Baseline; Metastatic 3rd Line | 10.2 [10.0 to 10.4]
  Change at Week 12; Adjuvant Chemotherapy: number analyzed (Participants) | 70
  Change at Week 12; Adjuvant Chemotherapy | 1.7 [1.4 to 2.0]
  Change at Week 12; Metastatic 1st or 2nd Line: number analyzed (Participants) | 92
  Change at Week 12; Metastatic 1st or 2nd Line | 1.6 [1.3 to 1.9]
  Change at Week 12; Metastatic 3rd Line: number analyzed (Participants) | 35
  Change at Week 12; Metastatic 3rd Line | 1.2 [0.8 to 1.7]

4. Secondary Outcome: Change From Baseline in Hemoglobin Levels After 12 Weeks of Study Treatment in Participants According to the Time Spent on Chemotherapy at Baseline
Description: Participants were distributed into 2 subgroups. One subgroup contained participants who had spent <6 months on chemotherapy and other subgroup contained participants who had spent 6 months or more on chemotherapy.
Time Frame: Baseline, Week 12
Population: Safety population. Here, "Number Analyzed" represents number of participants evaluable for the specified category.
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Epoetin Beta
Number analyzed (Participants) | 197
g/dL
  Baseline; <6 Months on Chemotherapy: number analyzed (Participants) | 152
  Baseline; <6 Months on Chemotherapy | 10.0 [9.9 to 10.1]
  Baseline; ≥6 Months on Chemotherapy: number analyzed (Participants) | 45
  Baseline; ≥6 Months on Chemotherapy | 10.0 [9.8 to 10.2]
  Change at Week 12; <6 Months on Chemotherapy: number analyzed (Participants) | 152
  Change at Week 12; <6 Months on Chemotherapy | 1.6 [1.4 to 1.8]
  Change at Week 12; ≥6 Months on Chemotherapy: number analyzed (Participants) | 45
  Change at Week 12; ≥6 Months on Chemotherapy | 1.4 [1.0 to 1.8]

5. Secondary Outcome: Overall Mean Change From Baseline in Hemoglobin Levels After 12 Weeks of Study Treatment
Time Frame: Baseline, Week 12
Population: Safety population
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Epoetin Beta
Number analyzed (Participants) | 197
g/dL
  Baseline | 10.0 [9.9 to 10.1]
  Change at Week 12 | 1.6 [1.4 to 1.8]

6. Secondary Outcome: Percentage of Participants With an Increase From Baseline in Hemoglobin Levels of At Least 1 g/dL After 4 Weeks
Time Frame: Baseline, Week 4
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Epoetin Beta
Number analyzed (Participants) | 197
percentage of participants | 45.4 [37.85 to 53.11]

7. Secondary Outcome: Mean Time Needed to Increase Hemoglobin Level by At Least 1 g/dL
Description: Time to increase in hemoglobin level by at least 1 g/dL was defined as the time between the start of treatment and an increase in hemoglobin level by at least 1 g/dL compared to baseline hemoglobin level. Time to response was estimated using Kaplan Meier method.
Time Frame: Baseline up to Week 12
Population: Safety population
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Epoetin Beta
Number analyzed (Participants) | 197
days | 34.2 [28 to 42]

8. Secondary Outcome: Quality of Life Assessment Using Functional Assessment of Cancer Therapy-Anemia (FACT-An) Questionnaire Scores
Description: FACT-An comprised of 2 subscales ('Fatigue' and 'Non-fatigue') of 20-items. All questions were rated on a scale from 0 to 4, where higher scores indicate improved quality of life. The 'Fatigue' subscale consists of 13 questions with score range from 0-52; 'Non-fatigue' subscale consists of 7 questions with score range from 0-28. Total FACT-An score was transformed to a 0-100 scale (instead of 0-80 scale) to get better perception of the participant's quality of life indicator.
Time Frame: Baseline, Week 12
Population: Safety population. Here, "Number of Participants Analyzed" represents number of participants evaluable for this outcome measure and "Number Analyzed" represents number of participants evaluable at specified time points.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Epoetin Beta
Number analyzed (Participants) | 162
units on a scale
  Baseline | 65.6 [63.2 to 67.9]
  Week 12: number analyzed (Participants) | 96
  Week 12 | 71.9 [68.6 to 75.2]

ADVERSE EVENTS:
Time Frame: Baseline up to Week 12
Description: Safety population
Arm/Group | Epoetin Beta
Serious Adverse Events (participants affected / at risk) | 17/197
Other Adverse Events (participants affected / at risk) | 85/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epoetin Beta (N=197)
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Disease progression (General disorders) | 2
Fatigue (General disorders) | 1
General physical health deterioration (General disorders) | 1
Contrast media reaction (Injury, poisoning and procedural complications) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Axillary vein thrombosis (Vascular disorders) | 1
Hypovolaemic shock (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Epoetin Beta (N=197)
Neutropenia (Blood and lymphatic system disorders) | 32
Leukopenia (Blood and lymphatic system disorders) | 18
Nausea (Gastrointestinal disorders) | 17
Asthenia (General disorders) | 32
Pyrexia (General disorders) | 17
Mucosal inflammation (General disorders) | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 15
Paraesthesia (Nervous system disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.